CLINICAL TRIAL: NCT06536023
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess Safety, Tolerability and Pharmacokinetics of IBI362 in Chinese Obese Adolescent Subjects
Brief Title: This is a Study to Evaluate the Pharmacokinetics and Safety of IBI362 in Chinese Adolescents With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362B103
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Adolescents With Obesity
MeSH Terms: interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 362-dose1-4mg (Experimental): The starting dose for the subjects is 2 mg, administered once weekly for 4 consecutive weeks. If the subject shows good tolerability, the dose will then be escalated to 4 mg, also given once weekly, for another 8 weeks (with an escalation rate of increasing 2 mg every 4 weeks until reaching the target dose).
  Interventions: Drug: IBI362
- 362-dose2-6mg (Experimental): Subjects start at a dose of 2 mg, administered once weekly for 4 consecutive weeks. Following this, if the subject demonstrates good tolerability#, the dose will be escalated to 4 mg, also administered once weekly, for another 4 weeks. After observing the subject's tolerability again, if it remains favorable#, the dose will be further escalated to 6 mg, administered once weekly, for another 4 weeks (dosing will increase by 2 mg every 4 weeks until reaching the target dose of 6 mg)
  Interventions: Drug: IBI362
- 362-dose3-Placebo (Experimental): Administration is via subcutaneous injection once weekly; the mode and form of placebo administration are consistent with those of IBI362, with continuous dosing over a 12-week period.
  Interventions: Drug: IBI362 placebo

INTERVENTIONS:
Drug: IBI362 — IBI362 SA.QW
  Arms: 362-dose1-4mg; 362-dose2-6mg
Drug: IBI362 placebo — IBI362 placebo SA.QW
  Arms: 362-dose3-Placebo

SUMMARY:
The study is a first-in-pediatric assessment of the safety, tolerability, and pharmacokinetic characteristics of multiple doses of IBI362 in Chinese adolescent subjects with obesity. It employs a multicenter, randomized, double-blind, and placebo-controlled trial design. The study plans to enroll 36 adolescents (aged ≥12 years and <18 years) with obesity who have experienced less than a 5% decrease in Body Mass Index (BMI) after at least 12 weeks of diet and exercise control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are aged ≥12 years and <18 years at the time of signing the informed consent;
2. At screening, the Body Mass Index (BMI) meets the obesity criteria according to "WS/T586-2018 Screening Criteria for Overweight and Obesity in School-age Children and Adolescents";
3. Subjects who have maintained a controlled diet and exercise for at least 12 weeks prior to screening, with no more than a 5% decrease in BMI (as reported by the subject, parent, or legal guardian);
4. Able to maintain a stable diet and exercise lifestyle during the study period;
5. Capable of understanding the procedures and methods of this study, willing to strictly adhere to the clinical trial protocol to complete this trial, with both the subject and the parent or legal guardian voluntarily signing the informed consent form.

Exclusion Criteria:

1. Prepubertal subjects (Tanner Stage I)
2. Subjects for whom the investigator suspects an allergy to the study drug or any of its components, or subjects with a history of allergies
3. Use of other weight-loss medications or treatments prior to screening
4. Evidence or history of other medical conditions prior to screening:

   * HbA1c ≥ 6.5% at screening or a previous diagnosis of Type 1 or Type 2 diabetes
   * Presence of retinopathy at screening
   * History of severe hypoglycemia or recurrent symptomatic hypoglycemia
   * Obesity secondary to disease or medication, including hypercortisolism (e.g., Cushing's syndrome)
   * Previous bariatric surgery
   * History of moderate to severe depression; or history of serious psychiatric illness
   * Previous suicidal ideation or suicide attempt

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | up to week 20

SECONDARY OUTCOMES:
Area under the Curve (AUC) of multi-dose of IBI362 | up to week 12
Half-life (t1/2) of multi-dose of IBI362 | up to week 12
Peak serum concentration (Cmax) of multi-dose of IBI362 | up to week 12
Clearance (CL) of multi-dose of IBI362 | up to week 12
Evaluate changes in subjects' fasting body weight in kilograms，Body Mass Index in kg/m2（BMI, combined with weight and height） relative to baseline | up to week 12
Evaluate changes in subjects' waist-to-hip ratio（combined with waistline and hips） relative to baseline | up to week 12
Evaluate changes in subjects' blood pressure in mmHg relative to baseline | up to week 12
Evaluate changes in subjects' lipid profile in mmol/L relative to baseline | up to week 12
Evaluate changes in subjects' glycated hemoglobin（Hemoglobin A1c,HbA1c）in % relative to baseline | up to week 12
Evaluate the mental health status of subjects by Patient Health Questionnaire (PHQ-9) following administration of IBI362. | up to week 20
Evaluate the mental health status of subjects by Columbia-Suicide Severity Rating Scale (C-SSRS) following administration of IBI362. | up to week 20

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Capital Medical University Affiliated, Beijin, Beijin, China

IPD SHARING:
Plan to Share IPD: No